CLINICAL TRIAL: NCT02530034
Title: Phase I Study of Hu8F4 in Patients With Advanced Hematologic Malignancies
Brief Title: Hu8F4 in Treating Patients With Advanced Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0057; NCI-2015-02131 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P-TRP-2447-14; 2014-0057 (Other: M D Anderson Cancer Center); P50CA100632 (NIH); NCI-2015-02131 (Other: NCI-CTRP Clinical Trials Reporting Registration)
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid Cell Neoplasm; High Risk Myelodysplastic Syndrome; Myelodysplastic Syndrome With Excess Blasts-1; Myelodysplastic Syndrome With Excess Blasts-2; Myelofibrosis; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Refractory Chronic Myelomonocytic Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Blast Crisis; Hematologic Neoplasms; Primary Myelofibrosis; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Hu8F4) (Experimental): Patients receive anti-PR1/HLA-A2 monoclonal antibody Hu8F4 IV over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-PR1/HLA-A2 Monoclonal Antibody Hu8F4; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Anti-PR1/HLA-A2 Monoclonal Antibody Hu8F4 — Given IV
  Other Names: Hu8F4
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of anti-PR1/HLA-A2 monoclonal antibody Hu8F4 (Hu8F4) in treating patients with malignancies related to the blood (hematologic). Monoclonal antibodies, such as Hu8F4, may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and minimum safe and biologically-effective dose of Hu8F4 when administered intravenously in patients with leukemia or myelodysplastic syndrome (MDS).

II. To determine the pharmacokinetics (PK) of Hu8F4 following study drug administration.

SECONDARY OBJECTIVES:

I. To observe the anti-leukemia effects of Hu8F4 in patients with leukemias and MDS.

II. To measure the overall survival, disease-free survival and event-free survival of patients with leukemias or MDS treated with Hu8F4.

OUTLINE: This is a dose-escalation study.

Patients receive anti-PR1/HLA-A2 monoclonal antibody Hu8F4 intravenously (IV) over 60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any of the following diagnoses are eligible: 1) high-risk MDS (i.e. refractory anemia with excess blasts [RAEB-1 or RAEB-2] by World Health Organization [WHO] classification, or any WHO subset with International Prognostic Scoring System [IPSS] intermediate-2 or high, or any patients that have failed prior therapy with hypomethylating agents); 2) chronic myelomonocytic leukemia (CMML); 3) acute myeloid leukemia (AML) by WHO classification; 4) chronic myeloid leukemia in blast phase (CML-BP); 5) myelofibrosis with high-risk features (e.g., accelerated phase disease -10-19% blasts in peripheral blood or bone marrow-, or with Dynamic International Prognostic Scoring System [DIPSS]-plus high risk score)
* Patients must have relapsed/refractory disease and have failed, or are not candidates for, or have declined all available therapies of proven efficacy; they should also not be eligible for at the time of enrollment or have declined hematopoietic stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* The effects of Hu8F4 on a fetus or nursing child are unknown; women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative urine pregnancy test within 2 weeks prior to beginning treatment on this trial; nursing patients are excluded; sexually active men must also use acceptable contraceptive methods for the duration of time on study
* Patients must have human leukocyte antigen (HLA)-A2 phenotype
* Must be able and willing to give written informed consent
* Patients must be at least 2 weeks from prior chemotherapy, radiation therapy, or major surgery, and at least 4 weeks or 5 half lives from other investigational anticancer therapy, and have recovered from prior toxicities at least to grade 1; the exception is hydroxyurea that requires no washout prior to the start of study drug
* Clinically significant toxicities from prior chemotherapy must not be greater than grade 1
* Clearance creatinine or glomerular filtration rate (GFR) >= 40 mL/min
* Total bilirubin =< 1.5 x the upper limit of normal unless considered due to Gilbert's syndrome or leukemic involvement
* Alanine aminotransferase (ALT) =< 3 x the upper limit of normal unless considered due to leukemic involvement

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to uncontrolled infection (patients must have no temperature >= 38.3 degrees Celsius [C] due to infection for at least 48 hrs to consider an infection controlled), psychiatric illness that would limit compliance with study requirements, or active heart disease including confirmed myocardial infarction within previous 3 months, symptomatic coronary artery disease, clinically significant arrhythmias not controlled by medication, or uncontrolled congestive heart failure New York (NY) Heart Association class III or IV
* Patients with current active malignancies or any remission for < 18 months, except patients with carcinoma in situ or with non-melanoma skin cancer who may have active disease or be in remission for less than 6 months
* Patients receiving any other standard or investigational treatment for their hematologic malignancy other than supportive care
* Patients who have had any major surgical procedure within 14 days of day 1
* Patients with known central nervous system infiltration with leukemia
* Patients who received an allogeneic stem cell transplant =< 90 days from the start of therapy
* Patients with active >= grade 3 graft versus host disease (GVHD), or receiving systemic steroids (> 10 mg/day of prednisone or equivalent) for GVHD
* Patients with known active central nervous system (CNS) disease; patients with history of active CNS disease should have at least two negative spinal fluid evaluations before being considered eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Minimum safety data | 4 weeks
  Safety data will be summarized using frequency and percentage for all patients.
Biologically-effective dose | 4 weeks
  Safety data will be summarized using frequency and percentage for all patients.

SECONDARY OUTCOMES:
Overall survival | Up to 4 years
  Estimated using the Kaplan-Meier methods.
Disease-free survival | Up to 4 years
  Estimated using the Kaplan-Meier methods.
Event-free survival | Up to 4 years
  Estimated using the Kaplan-Meier methods.
Duration of complete remission | Up to 4 years
  Complete remission rates will be estimated along with 95% credible intervals. Estimated using the Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Augusta University, Augusta, Georgia
  - Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org